CLINICAL TRIAL: NCT04655794
Title: Clinical Analysis of Safety in Latent Tuberculosis Infection Prophylaxis Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201800081B0
Record Dates: First submitted 2020-11-24; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Adverse Reaction to Drug; 3HP
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- had >= grade 2 adverse reactions
  Interventions: Drug: 3HP
- had <2 frade 2 adverse reactions
  Interventions: Drug: 3HP

INTERVENTIONS:
Drug: 3HP — all patients taking 3HP under directly observed preventive therapy (DOPT) program

SUMMARY:
The treatment of latent TB with 3HP is an important issue for the prevention of active TB. However, significant proportion of subjects receiving 3HP had adverse reaction. The main purpose of this observation study is to identify subjects who have higher risk to develop adverse reaction. Clinical characteristics and biomarker will be used to predict adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

* close contact with active TB patients
* patients with autoimmune diseases preceding biological therapy
* health-care workers
* other clinical conditions, which increased the risk of LTBI. LTBI was confirmed by QuantiFERON-TB Gold In-Tube test (QFT-GIT; Qiagen, Valencia, CA, USA) with a cut-off value of 0.35 IU/ml.

Exclusion Criteria:

* age less than 20 years
* pregnant women
* active TB or suspected active TB in the clinical evaluation
* severe liver disease
* ESRD
* organ transplantation
* close contact with a multidrug-resistant TB patient
* obesity (BMI>30 Kgw/m2) and other conditions inappropriate for participation in this study as judged by the investigators.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The newly identified LTBI subjects who wanted to receive LTBI preventive therapy with 3HP were eligible for enrolment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-02-12 (Estimated)

PRIMARY OUTCOMES:
sTREM1 between >= grade 2 adverse reaction (SAR group) and< grade 2 adverse reaction (Non-SAR group) | Change from Baseline sTREM1 at 2 weeks
sTREM1 between >= grade 2 adverse reaction (SAR group) and< grade 2 adverse reaction (Non-SAR group) | Change from Baseline sTREM1 at SARs
sTREM2 between >= grade 2 adverse reaction (SAR group) and< grade 2 adverse reaction (Non-SAR group) | Change from Baseline sTREM1 at 2 weeks
sTREM2 between >= grade 2 adverse reaction (SAR group) and< grade 2 adverse reaction (Non-SAR group) | Change from Baseline sTREM1 at SARs

CONTACTS AND LOCATIONS:
Locations (1):
- Institutional Review Board Chang Gung Medical Foundation, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang TY, Feng JY, Shu CC, Lee SS, Chen CY, Wei YF, Lin CB, Huang WC, Su WJ, Lin SM. Plasma Concentrations of sTREM-1 as Markers for Systemic Adverse Reactions in Subjects Treated With Weekly Rifapentine and Isoniazid for Latent Tuberculosis Infection. Front Microbiol. 2022 Mar 3;13:821066. doi: 10.3389/fmicb.2022.821066. eCollection 2022. PMID 35308376